CLINICAL TRIAL: NCT04478539
Title: Clinical Efficacy and Safety of Extracorporeal Blood Purification to Control Hyperinflammation and Hypercoagulability in COVID-19 Patients
Brief Title: Extracorporeal Blood Purification as a Treatment Modality for COVID-19
Status: Completed | Type: Observational
Sponsor: Zan Mitrev Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: EBPZ.357
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2; cytokine storm; Interleukin 6; hypercoagulability; Fibrinogen; D-dimer
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- COVID-19 patients admitted to the ICU: COVID-19 patients will be treated with the Prismaflex® oXiris® system in the ICU.
  Treatment will be initiated within 4 - 12 hours after admission upon establishing control of the haemostasis, ACT = Activated Coagulation Time of 180 seconds
  Interventions: Device: Extracorporeal blood purification using the oXiris® (AN69ST) hemofilter

INTERVENTIONS:
Device: Extracorporeal blood purification using the oXiris® (AN69ST) hemofilter — Admitted patients will receive at least 1 cycle of extracorporeal blood purification using the oXiris® (AN69ST) hemofilter (Baxter, IL, USA). The number of cycles of blood purification is determined based on multiple biochemical, immunological, coagulation parameters, radiological imaging and overall clinical condition.
  The patient is connected to the Prismaflex® oXiris® system via a double lumen catheter placed in the femoral vein or vena subclavia.
  Flow rates will be maintained as follow; effluent dose 35 mL/Kg/h, dialysate 14 - 16 mL/Kg/h, blood 150 mL/min, replacement 16 -18 mL/Kg/h; patient fluid removal is tailored to the individual's volume status, ≈ 100 - 250 mL/h.
  The oXiris® extracorporeal and organ support modality will be chosen according to the patient's kidney function; continuous venovenous hemofiltration (CVVH), continuous venovenous hemodiafiltration (CVVHDF) or slow continuous ultrafiltration (SCUF).

SUMMARY:
Several studies have suggested a potential clinical benefit of controlling hyper inflammation triggered by SARS-CoV-2/COVID-19. Blood purification, the removal of excessive proinflammatory mediators may control disease progression and support clinical recovery.

For this purpose, COVID-19 patients might benefit from treatment with AN69ST hemofilter based extracorporeal blood purification.

DETAILED DESCRIPTION:
COVID-19 disease progression is associated with dysregulated immunity, commonly referred to as cytokine storm, in particular, aberrant Interleukin (IL) 6 levels that promote numerous pathological downstream effects. Hyperinflammation is a well-established trigger of multiorgan failure, for example, acute kidney injury. Moreover, recent reports point to a link between hyper inflammation and COVID-19 induced coagulopathy as a result of increased production of clotting factors by the liver.

Despite several lines of evidence pointing to a potential clinical benefit of controlling hyperinflammation triggered by COVID-19, management of COVID-19 remains mostly supportive built around continuous respiratory support.

To this end, considering the underlying immunological character of COVID-19 disease and the high risk of SARS-CoV-2 hyperinflammation to trigger ARDS, hypercoagulability and Acute Kidney Injury (AKI) this study aims to monitor selected biochemical, immunological and coagulation parameters in combination with radiological imaging to guide clinical practice and to tailor therapy consisting of 1) early initiation of blood purification using the oXiris® (AN69ST) filter, 2) systemic heparinisation and 3) respiratory support

ELIGIBILITY:
Inclusion Criteria:

Confirmed COVID-19 disease:

* RT-PCR
* Atypical Pneumonia; X-Ray and/or Computed Tomography
* ≥ 1 oXiris® blood purification cycle

Exclusion Criteria:

* Pregnancy
* Heart failure; severe systolic dysfunction, left ventricular ejection fraction < 25% requiring urgent surgery
* Aortic Aneurysms, dissection or rupture requiring urgent surgery
* Recent Myocardial Infarction; cardiovascular disease patients requiring urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID positive patients admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in cytokine levels of Interleukin (IL) 6, IL-8 and Tumor Necrosis Factor-α (pg/mL) | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Systemic levels of IL-6, IL-8 and TNF-α are evaluated to assess the effect of blood purification.
  Measurement points: at admission, "before and after a blood purification cycle" and before discharge
Changes in inflammatory markers; C-Reactive Protein (CRP) (mg/L) | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Systemic levels of proinflammatory mediators are measured as a marker for disease severity.
  Measurement points: at admission, "before and after a blood purification cycle" and before discharge.
Changes in thrombocyte counts (10^3 counts/microL) | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Systemic levels of thrombocytes are measured as a marker for disease severity.
  Measurement points: at admission, "before and after a blood purification cycle" and before discharge.
Changes in the coagulation marker Fibrinogen (g/L) | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Coagulation markers will be followed to assess the effect of systemic heparinisation,
  Measurement points, at admission, "before and after a blood purification cycle" and before discharge
ICU length of stay after admission (days) | An expected average of 4 - 14 hospitalisation days or until hospital discharge (whichever comes first)
  Duration of intensive care will be determined in relation to the number of blood purification cycles
  Patients will be followed for the duration of ICU stay.

SECONDARY OUTCOMES:
Changes in Neutrophil-to-Lymphocyte Ratio | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Systemic levels of proinflammatory mediators are measured as a marker for disease severity.
  Measurement points: at admission, "before and after a blood purification cycle" and before discharge.
Changes in the coagulation marker D-Dimers (ng/mL) | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Coagulation markers will be followed to assess the effect of systemic heparinisation,
  Measurement points, at admission, "before and after a blood purification cycle" and before discharge
Changes in the Activation Clotting Time (seconds). | Hospitalisation window, day 0 until day 14 or until hospital discharge (whichever comes first)
  Coagulation markers will be followed to assess the effect of systemic heparinisation,
  Measurement points, at admission, "before and after a blood purification cycle" and before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Zan K Mitrev, MD, Study Director — Zan Mitrev Clinic; Rodney A Rosalia, PhD, Principal Investigator — Zan Mitrev Clinic
Locations (1):
- Zan Mitrev Clinic, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malard B, Lambert C, Kellum JA. In vitro comparison of the adsorption of inflammatory mediators by blood purification devices. Intensive Care Med Exp. 2018 May 4;6(1):12. doi: 10.1186/s40635-018-0177-2. PMID 29728790
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] The Lancet Haematology. COVID-19 coagulopathy: an evolving story. Lancet Haematol. 2020 Jun;7(6):e425. doi: 10.1016/S2352-3026(20)30151-4. No abstract available. PMID 32470428
- [Background] Herold T, Jurinovic V, Arnreich C, Lipworth BJ, Hellmuth JC, von Bergwelt-Baildon M, Klein M, Weinberger T. Elevated levels of IL-6 and CRP predict the need for mechanical ventilation in COVID-19. J Allergy Clin Immunol. 2020 Jul;146(1):128-136.e4. doi: 10.1016/j.jaci.2020.05.008. Epub 2020 May 18. PMID 32425269
- [Background] Zhang Y, Yu L, Tang L, Zhu M, Jin Y, Wang Z, Li L. A Promising Anti-Cytokine-Storm Targeted Therapy for COVID-19: The Artificial-Liver Blood-Purification System. Engineering (Beijing). 2021 Jan;7(1):11-13. doi: 10.1016/j.eng.2020.03.006. Epub 2020 Mar 20. No abstract available. PMID 32292628
- See also: FDA Emergency Use Authorization for Oxiris Blood Purification Filter for COVID-19 Treatment — https://www.baxter.com/baxter-newsroom/baxter-obtains-us-fda-emergency-use-authorization-oxiris-blood-purification-filter